CLINICAL TRIAL: NCT00548899
Title: Phase II Study of Neoadjuvant Epirubicin, Cyclophosphamide (EC) + Sorafenib Followed by Paclitaxel (P) + Sorafenib in Women With Previously Untreated
Brief Title: Neoadjuvant Chemotherapy Including Sorafenib in Women With Previously Untreated Primary Breast Cancer
Acronym: SOFIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBG 45; 2007-000124-41 (EudraCT Number)
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant chemotherapy; Targeted therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Other): Single Arm: All patients receive sorafenib in addition to the established chemotherapy
  Interventions: Drug: Nexavar (Sorafenib)

INTERVENTIONS:
Drug: Nexavar (Sorafenib) — Tablet, Sorafenib follows a patient specific escalation scheme starting with 200 mg daily up to a maximum dose of 800 mg daily during EC chemotherapy on day 2-19. The achieved dose will be continued during paclitaxel chemotherapy during week 1-11 all day

SUMMARY:
The purpose of this study is to determine the efficacy and safety of sorafenib in the neoadjuvant setting in patients with primary breast cancer

DETAILED DESCRIPTION:
Epirubicin/Cyclophosphamide followed by Paclitaxel (EC/P) is a well tolerated regimen with high clinical activity. Histopathological complete remission after preoperative chemotherapy has a direct correlation with the disease-free and overall survival. The aim of combining a chemotherapy regime with sorafenib in the neoadjuvant setting is to increase the locoregional and systemic outcome of these patients

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral primary carcinoma of the breast,
* Tumor lesion in the breast with a palpable size of >= 2 cm. The lesion has to be measurable in two-dimensions preferably by sonography. In case of inflammatory disease the extent of inflammation can be used as measurable lesion;
* Patients should have stages of disease in which adjuvant chemotherapy would be considered.
* Women of childbearing potential must have a negative serum pregnancy test
* Negative HER-2/neu status
* Karnofsky Performance status index >= 80%;
* Normal cardiac function
* Laboratory requirements:

Absolute neutrophile count (ANC) >= 2,0 x 109/L and Platelets >= 100 x 109/L and Hemoglobin >= 10 g/dL (>= 6.2 mmol/L) INR ≤ 1.5 ULN and PTT ≤ 1.5 ULN within 14 days prior to enrolment ASAT or ALAT < 2.5 x ULN Alkaline phosphatase ≤ 5 UNL. Patients with ASAT and/or ALAT > 1,5 x UNL associated with alkaline phosphatase > 2,5 x UNL are not eligible for the study Total bilirubin < 1 X UNL Creatinine ≤ 175 µmol/L (2 mg/dl). The calculated creatinine clearance should be ≥ 60 mL/min.

Paraffin tumor tissue block and each one serum and one plasma sample centrally made available

* Complete staging work-up within 3 months prior to registration.
* Patients must be available and compliant for treatment and follow-up. Patients registered on this trial must be treated and followed up at the participating or a cooperating center.

Exclusion Criteria:

* Patients with low or moderate risk, which are only doubtful candidates for adjuvant chemotherapy and do not fulfil the inclusion criteria No. 5.
* Evidence of distant metastasis;
* Prior chemotherapy for any malignancy;
* Prior radiation therapy for breast cancer;
* Preexisting rhagades at hand and feet and other skin problems (e.g. psoriasis)
* Pregnant or lactating patients.
* Pre-existing motor or sensory neuropathy of a severity >= grade 2 by NCI criteria; 7. Concurrent treatment with: Chronic corticosteroids unless initiated > 6 months prior to study entry and at low dose (< 20 mg methylprednisolone or equivalent); Sex hormones. Prior treatment must be stopped before study entry; Patients with increased risk of bleeding due to concurrent therapeutic or prophylactic anticoagulative treatment. Low dose of coumarines are permitted.

Other experimental drugs or any other anti-cancer therapy; Drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A within the last 5 days or their expected need 8. Other serious illness or medical condition:

* Previous malignant disease without being disease-free of less than 5 years (except CIS of the Cervix and non-melanomatous skin cancer)
* Known or suspected congestive heart failure (≥NYHA II) and/or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, un- or poorly controlled arterial hypertension, rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease
* Thrombotic or embolic events
* Hemorrhage/bleeding event ≥ Grade 3 within 4 weeks prior study entry
* Evidence or history of bleeding diathesis or coagulopathy
* History of significant neurological or psychiatric disorders
* Patients with seizure disorders requiring medication such as steroids or antiepileptics
* Currently active infection
* History of HIV infection or chronic hepatitis B or C
* Serious non healing wound, ulcer or bone fracture
* Patients with prior immunosuppressive treatment
* Severe pulmonary condition/illness
* Disease significantly affecting gastrointestinal function,
* Patients with severe liver disease
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first dose of study drug
* Definite contraindications for the use of corticosteroids
* Inadequate general condition (not fit for anthracycline/taxane-containing chemotherapy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-11; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
to establish the most feasible regimen of EC-P (P-EC) with sorafenib | Time of surgery

SECONDARY OUTCOMES:
Safety of preoperative regimen | Treatment to Surgery
Determine clinical response rate | Time of surgery
Histopathological axillary nodal status after neoadjuvant therapy | Time of surgery
Correlate baseline and change in tumor and serum genetic, gene expression and proteomic patterns with clinical and pathological response | Baeline till time of surgery
pCR rate at surgery | Treatment ot Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Loibl, MD, Study Chair — GBG Forschungs GmbH
Locations (9):
- Germany (9):
  - St. Gertrauden Krankenhaus, Berlin
  - Klinikum der Universität zu Köln, Cologne
  - Klinikum der J. W. Goethe Universität, Frankfurt am Main
  - Henriettenstiftung, Hanover
  - Elisabeth Krankenhaus, Kassel
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Klinikum Offenbach, Offenbach
  - Klinikum Südstadt, Rostock
  - Dr.-Horst-Schmidt-Kliniken GmbH, Wiesbaden

REFERENCES:
- [Result] Loibl S, Rokitta D, Conrad B, Harbeck N, Wullner M, Warm M, Schwedler K, Gerber B, Schrader I, Eidtmann H, Mehta K, Fuhr U, von Minckwitz G. Sorafenib in the Treatment of Early Breast Cancer: Results of the Neoadjuvant Phase II Study - SOFIA. Breast Care (Basel). 2014 Jul;9(3):169-74. doi: 10.1159/000363430. PMID 25177258
- See also: Related Info — http://www.germanbreastgroup.de